CLINICAL TRIAL: NCT01759329
Title: Health Effects of Coffee Consumption
Acronym: DüsselKaffee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Collaborators: Tchibo GmbH (Unknown)
Responsible Party: Principal Investigator, Stephan Martin, principal investigator, West German Center of Diabetes and Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DüsselKaffee
Record Dates: First submitted 2012-12-21; First posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Overweight
Keywords: overweight; body weight; coffee
MeSH Terms: conditions — Overweight; Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- test coffee (Experimental): test coffee
  Interventions: Dietary Supplement: test coffee
- control coffee (Active Comparator): control coffee
  Interventions: Dietary Supplement: control coffee

INTERVENTIONS:
Dietary Supplement: test coffee — test coffee with higher alkyl pyridine content
  Arms: test coffee
Dietary Supplement: control coffee — control coffee with regular alkyl pyridine content
  Arms: control coffee

SUMMARY:
Epidemiological studies have indicated a positive health impact of coffee. Nevertheless, intervention studies testing the effect of daily coffee consumption over a longer period are lacking so far. Moreover, there is a lack of knowledge about the properties of different coffees and their influence on weight development. Therefore, we tested the effect of two coffees differing in their alkyl pyridine content over a period of 3 months on weight development.

DETAILED DESCRIPTION:
Participants were randomly associated to two groups, a test coffee group and a control coffee group. After coffee abstinence of 1 months, participants in both groups got a coffee machine and coffee pads for three months. Clinical data have been assessed before and after coffee abstinence and after 3 months of coffee consumption.

ELIGIBILITY:
Inclusion Criteria:

* age 18-69 years
* BMI ≥27 kg/m2
* coffee consumption of ≥3 cups per day

Exclusion Criteria:

* new diagnosed type 2 diabetes during the last 6 months
* severe diseases with hospital stay during the last 3 months
* change of body weight of more than 2 kg per week during the last 4 weeks
* smoking cessation during the last 3 months or planned during the study
* acute infects
* chronical diseases with except of type 2 diabetes mellitus
* regular pharmacological therapy with except of oral antidiabetic medication or contraception
* lack of contraception in women
* breastfeeding
* physical activity of more than 1 hour per day

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
body weight | 4 months
  body weight

CONTACTS AND LOCATIONS:
Overall Officials: Stepahn Martin, MD, Principal Investigator — WDGZ
Locations (1):
- West German Center of Diabetes and Health, Düsseldorf, Germany

REFERENCES:
- [Derived] Kempf K, Kolb H, Gartner B, Bytof G, Stiebitz H, Lantz I, Lang R, Hofmann T, Martin S. Cardiometabolic effects of two coffee blends differing in content for major constituents in overweight adults: a randomized controlled trial. Eur J Nutr. 2015 Aug;54(5):845-54. doi: 10.1007/s00394-014-0763-3. Epub 2014 Sep 10. PMID 25204719